CLINICAL TRIAL: NCT00332579
Title: A Double-Blind, Placebo-Controlled Study of Naltrexone in Kleptomania
Brief Title: Double-Blind Naltrexone in Kleptomania
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0602M82626
Record Dates: First submitted 2006-05-30; First posted 2006-06-01 (Estimated); Results first posted 2012-05-04 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Kleptomania
Keywords: Compulsive Shoplifting; Kleptomania; Compulsive Stealing
MeSH Terms: conditions — Disruptive, Impulse Control, and Conduct Disorders | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Naltrexone
  Interventions: Drug: Naltrexone
- B (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — daily
  Other Names: Revia
  Arms: A
Drug: Placebo — daily
  Arms: B

SUMMARY:
The goal of the proposed study is to evaluate the efficacy and safety of naltrexone in kleptomania.

DETAILED DESCRIPTION:
The proposed study will consist of 8 weeks of treatment with either naltrexone or placebo in 20 subjects with kleptomania. The hypothesis to be tested is that naltrexone will be effective in reducing the urges to steal in patients with kleptomania. The proposed study will provide needed data on the treatment of a disabling disorder that currently lacks a clearly effective treatment.

ELIGIBILITY:
Inclusion Criteria:

1. men and women age 21-75
2. current DSM-IV kleptomania.

Exclusion Criteria:

1. unstable medical illness or clinically significant abnormalities on prestudy laboratory tests or physical examination
2. history of seizures
3. myocardial infarction within 6 months
4. current pregnancy or lactation, or inadequate contraception in women of childbearing potential
5. clinically significant suicidality
6. current or recent (past 3 months) DSM-IV substance abuse or dependence
7. illegal substance within 2 weeks of study initiation
8. initiation of psychotherapy or behavior therapy from a mental health professional for the treatment of kleptomania within 3 months prior to study baseline
9. initiation of a psychotropic medication within 2 months prior to study inclusion
10. previous treatment with naltrexone
11. treatment with investigational medication or depot neuroleptics within 3 months, with fluoxetine within 6 weeks, or with other psychotropics within 2 weeks prior to study baseline.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-05-01 (Actual); Primary Completion 2008-09-01 (Actual); Study Completion 2008-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, MD, JD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Grant JE, Kim SW, Odlaug BL. A double-blind, placebo-controlled study of the opiate antagonist, naltrexone, in the treatment of kleptomania. Biol Psychiatry. 2009 Apr 1;65(7):600-6. doi: 10.1016/j.biopsych.2008.11.022. Epub 2009 Feb 12. PMID 19217077

RESULTS

PARTICIPANT FLOW:
Groups:
- Naltrexone: Naltrexone 50mg tablets taken daily. Dose range from 50mg-150mg by mouth daily. Started at 50mg and then titrated up based upon investigator discretion.
- Placebo: Placebo tablets (identical to naltrexone pills) taken by mouth daily.
Period: Overall Study
Arm/Group | Naltrexone | Placebo
Started | 12 | 13
Completed | 11 | 12
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone | Placebo | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 13 | 25
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (12.2) | 41.4 (12.7) | 42.6 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Yale Brown Obsessive Compulsive Scale Modified for Kleptomania (K-YBOCS)
Description: The K-YBOCS measures symptom severity (urges/thoughts and behavior) across the past week. Scores range from 0 (no symptoms) to 40 (highest symptom severity).
Time Frame: K-YBOCS is done at each visit by the investigator.
Population: Reported scores are Mean and standard deviation for Subjects last visit (Week 8 or last-observation carried forward).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 12 | 13
units on a scale | 3.83 (2.86) | 11.46 (7.76)

ADVERSE EVENTS:
Arm/Group | Naltrexone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 5/13 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone (N=13) | Placebo (N=12)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Insomnia (General disorders) | 1 (1) | 0 (0)
Dry Mouth (General disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No